CLINICAL TRIAL: NCT02602093
Title: (Cost) Effectiveness of Percutaneous Transforaminal Endoscopic Discectomy vs. Open Microdiscectomy for Patients With Symptomatic Lumbar Disc Herniation
Brief Title: Percutaneous Transforaminal Endoscopic Discectomy vs. Open Microdiscectomy for Lumbar Disc Herniation (PTED-study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); VU University of Amsterdam (Other); Erasmus Medical Center (Other); The Elisabeth-TweeSteden Hospital (Other); Rijnstate Hospital (Other); Alrijne Hospital (Other); Park MC (Unknown)
Responsible Party: Principal Investigator, P.S. Gadjradj, MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZonMw 80-83700-98-15503
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disk Herniation
Keywords: Lumbar Disk Herniation; Percutaneous Transforaminal Endoscopic Discectomy; Micro Discectomy; Minimal Invasive Spine Surgery
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transforaminal Endoscopic Discectomy (Active Comparator): Surgery: Patients will undergo Percutaneous Transforaminal Endoscopic Discectomy.
  Interventions: Procedure: Transforaminal Endoscopic Discectomy
- Open Microdiscectomy (Active Comparator): Surgery: Patients will undergo conventional micro discectomy.
  Interventions: Procedure: Open Microdiscectomy

INTERVENTIONS:
Procedure: Transforaminal Endoscopic Discectomy — Local anaesthesia is to be administered. Verification of the site to be performed by an image intensifier and depending upon the patient's posture, a line is to be drawn from the center of the herniation. The needle is to be set and position checked. After the needle has reached the correct position, a guidewire is inserted. Following that, a series of conical rods are introduced, subsequently a drill is introduced through the cannula. After drilling, the instruments are removed, but the guidewire is to remain in place. The endoscope with the working channels are introduced via an 8mm cannula. Following removal of the hernia, the cannula and endoscope are removed. The patient is to be treated on an outpatient basis.
  Other Names: PTED
  Arms: Transforaminal Endoscopic Discectomy
Procedure: Open Microdiscectomy — General or spinal anaesthesia is to be administered. Verification is to be performed using a Carm and the patient is to be positioned prone or in the salaam position. A paramedian incision is to be performed and the level is to be indicated. Loupe or microscope magnification is to be used. Laminotomy as well as foraminotomy is to be performed, if necessary. The amount of degenerative disc material to be removed is at the discretion of the attending surgeon. Post-operative policy will be followed and it is expected that the duration of recovery in the hospital may vary from 2-7 days, but the patient will be discharged as soon as medically responsible.
  Other Names: OM
  Arms: Open Microdiscectomy

SUMMARY:
Rationale: Lumbosacral radicular syndrome (LSRS) is caused by a herniated lumbar nucleus pulposus (HNP) and the estimated annual incidence in The Netherlands ranges between 60,000 to 75,000 people. Open microdiscectomy is the standard surgical technique.

In recent years, several surgical techniques have been developed including, percutaneous transforaminal endoscopic discectomy (PTED). While PTED is gaining popularity in The Netherlands, evidence of its effects is lacking, leading to a heated debate. The current position of Zorginstituut Nederland (ZiN) is that there is insufficient evidence to support its use; therefore, PTED is not financially covered. The consequence is, patients are forced to pay the costs of treatment themselves. This study is expected to provide the necessary data to answer the question regarding effects and costs of PTED vs. open microdiscectomy, and help resolve the current debate.

DETAILED DESCRIPTION:
Rationale: Lumbosacral radicular syndrome (LSRS) is caused by a herniated lumbar nucleus pulposus (HNP) and the estimated annual incidence in The Netherlands ranges between 60,000 to 75,000 people. Open microdiscectomy is the standard surgical technique.

In recent years, several surgical techniques have been developed including, percutaneous transforaminal endoscopic discectomy (PTED). While PTED is gaining popularity in The Netherlands, evidence of its effects is lacking, leading to a heated debate. The current position of Zorginstituut Nederland (ZiN) is that there is insufficient evidence to support its use; therefore, PTED is not financially covered. The consequence is, patients are forced to pay the costs of treatment themselves. This study is expected to provide the necessary data to answer the question regarding effects and costs of PTED vs. open microdiscectomy, and help resolve the current debate. Objective: To determine the effects and costs of PTED vs. open microdiscectomy. Study design: Pragmatic, multi-center non-inferiority randomized controlled trial (RCT) with subsequent observational study once sufficient subjects have been recruited for the RCT.

Study population: In total, 682 subjects are to be included, with including 50 patients in the PTED-group per surgeon who will learn the procedure "the learning curve". Therefore, for the 3 surgeons who will learn the technique, the first 50 patients who will undergo PTED (150 total) will be analyzed seperatly.

The inclusion criteria are as follows: subjects 18-70 years of age with > 10 weeks of radiating pain with- or without motor or sensory loss in the leg, or with > 6 weeks of excessive radiating pain and no tendency for any clinical improvement and strong patient preference for surgery. There must also be an indication for an operation and a MRI demonstrating lumbar disc herniation with nerve compression with or without concomitant spinal or lateral recess stenosis or sequestration.

Participants must also have sufficient knowledge of the Dutch language.

ELIGIBILITY:
Inclusion Criteria:

* 10 weeks of radiating pain with- or without motor or sensory loss in the leg, or with > 6weeks of excessive radiating pain and no tendency for any clinical improvement and strong patient preference for surgery;
* Indication for an operation according to consensus;
* MRI demonstrating lumbar disc herniation with nerve compression with or without concomitant spinal or lateral recess stenosis or sequestration;
* Sufficient knowledge of the Dutch language in order to complete forms and follow instructions independently.

Exclusion Criteria:

* Previous surgery on the same or adjacent disc level;
* Cauda equina syndrome (CES);
* Spondylytic or degenerative spondylolisthesis;
* Pregnancy;
* Severe comorbid medical or psychiatric disorder (ASA>2);
* Severe caudal or cranial sequestration;
* Moving abroad at short notice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes on the Visual Analogue Scale for Leg Pain | Baseline, Day after surgery, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12, 24 and 60 months after surgery NRS was added for internal validation
  The pain intensity in the leg will be measured on a scale from 0 to 100 mm

SECONDARY OUTCOMES:
Changes on the Oswestry Disability Index | Baseline, Day after surgery, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months , 12, 24 and 60 months after surgery
  There are 10 questions (items), each with 6 possible answers, each answer option receives a score of 0 to 5 points, yielding score range between 0 and 50, which is scaled to a 100% range. The questions are designed in a way to realize how the back or leg pain is affecting the patient's ability to manage in everyday life
Costs of treatment measured using cost questionnaires filled out by the patients | Baseline, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months and , 12 and 24 months after surgery
  Cost questionnaires will be completed at the prescribed measurements. Hospitalisation for surgery will be registered using the case record forms. Other health care utilization (including physiotherapy, visits to GP and specialists, nursing care and medication), patient costs, and absenteeism from work will be measured using cost questionnaires filled out by the patients.
Changes on the Visual Analogue Scale for Back Pain | Baseline, Day after surgery, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12, 24 and 60 months after surgery NRS was added for internal validation
  The pain intensity in the back will be measured on a scale from 0 (no pain) to 100 mm (worst imaginable pain). An NRS was added as well.
Changes on the Quality of Life Visual Analogue Scale. | Baseline, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12, 24 and 60 months after surgery. NRS was added for internal validation
  To represent the patients' perspective, utility will also be estimated using a VAS for the valuation of the patient's health state (ranging from 0 = as bad as death to 100 mm = perfect health). An NRS was added as well.
Changes on the EuroQoL (EQ-5D) | Baseline, Day after surgery, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12 and 24 months after surgery
  The EuroQoL (EQ-5D) will be used for the cost utility analysis. The tool measures five dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each dimension consists of one item, while five levels are distinguished (no, slight, moderate, severe problems, unable to do).
Perceived recovery | Day after surgery, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12, 24 and 60 months after surgery
  To measure the perceived recovery a seven-point Likert scale will be used. The score on this scale vary from 'completely recovered' to 'worse than ever'.
Patient satisfaction | 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12, 24 and 60 months after surgery
  To measure patient satisfaction a seven-point Likert scale will be used. The score on this scale vary from 'completely satisfied with current symptoms' to 'completely dissatisfied with current symptoms'.
Changes on the SF-36 | Baseline, 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 9 months, 12, 24 and 60 months after surgery
  The SF-36 will be used as a generic quality-of-life questionnaire. The SF-36 questionnaire has been validated and found reliable for low back pain.
Complications | through study completion, up to 1, 2 year and 5 of follow-up
  A systematic assessment of complications (including wound infection, deep venous thrombosis, urine tract infection, hematoma, and progressive neurological deficit) will be recorded out by the surgeon and research nurse, and these data are to be extracted from the patient chart. Moreover, surgeons will be asked for perioperative complications
Physical Examination | Baseline, 6 weeks, 3 months and 12 months after surgery
  The wound will be inspected and a standard neurological examination will be performed. This standard neurologic examination includes the Body Image and Cosmesis Scale, the (crossed) leg raising test, patellar and tendon reflexes, sensibility in the lumbosacral dermatome region, leg muscle test, abdominal muscle strength and finger-floor distance.

CONTACTS AND LOCATIONS:
Overall Officials: Biswadjiet Harhangi, MD, PhD, Study Director — Erasmus Medical Center; Sidney Rubinstein, PhD, Principal Investigator — VU
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 24 months
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Seiger A, Gadjradj PS, Harhangi BS, van Susante JL, Peul WC, van Tulder MW, de Boer MR, Rubinstein SM. PTED study: design of a non-inferiority, randomised controlled trial to compare the effectiveness and cost-effectiveness of percutaneous transforaminal endoscopic discectomy (PTED) versus open microdiscectomy for patients with a symptomatic lumbar disc herniation. BMJ Open. 2017 Dec 21;7(12):e018230. doi: 10.1136/bmjopen-2017-018230. PMID 29273659
- [Background] Gadjradj PS, Harhangi BS. Percutaneous Transforaminal Endoscopic Discectomy for Lumbar Disk Herniation. Clin Spine Surg. 2016 Nov;29(9):368-371. doi: 10.1097/BSD.0000000000000366. PMID 26945128
- [Background] Gadjradj PS, van Tulder MW, Dirven CM, Peul WC, Harhangi BS. Clinical outcomes after percutaneous transforaminal endoscopic discectomy for lumbar disc herniation: a prospective case series. Neurosurg Focus. 2016 Feb;40(2):E3. doi: 10.3171/2015.10.FOCUS15484. PMID 26828884
- [Background] Gadjradj PS, Depauw PR, Schutte PJ, Vreeling AW, Harhangi BS. Body Image and Cosmesis after Percutaneous Transforaminal Endoscopic Discectomy versus Conventional Open Microdiscectomy for Sciatica. Global Spine J. 2024 Mar;14(2):390-399. doi: 10.1177/21925682221105271. Epub 2022 May 24. PMID 35610755
- [Background] Gadjradj PS. Full-endoscopic lumbar disc surgery: the new gold standard? (PhD Academy Award). Br J Sports Med. 2022 May 19:bjsports-2022-105434. doi: 10.1136/bjsports-2022-105434. Online ahead of print. No abstract available. PMID 35589376
- [Background] Gadjradj PS, Rubinstein SM, Peul WC, Depauw PR, Vleggeert-Lankamp CL, Seiger A, van Susante JL, de Boer MR, van Tulder MW, Harhangi BS. Full endoscopic versus open discectomy for sciatica: randomised controlled non-inferiority trial. BMJ. 2022 Feb 21;376:e065846. doi: 10.1136/bmj-2021-065846. PMID 35190388
- [Background] Gadjradj PS, Broulikova HM, van Dongen JM, Rubinstein SM, Depauw PR, Vleggeert C, Seiger A, Peul WC, van Susante JL, van Tulder MW, Harhangi BS. Cost-effectiveness of full endoscopic versus open discectomy for sciatica. Br J Sports Med. 2022 Feb 20;56(18):1018-25. doi: 10.1136/bjsports-2021-104808. Online ahead of print. PMID 35185010
- [Background] Gadjradj PS, Harhangi BS, Amelink J, van Susante J, Kamper S, van Tulder M, Peul WC, Vleggeert-Lankamp C, Rubinstein SM. Percutaneous Transforaminal Endoscopic Discectomy Versus Open Microdiscectomy for Lumbar Disc Herniation: A Systematic Review and Meta-analysis. Spine (Phila Pa 1976). 2021 Apr 15;46(8):538-549. doi: 10.1097/BRS.0000000000003843. PMID 33290374